CLINICAL TRIAL: NCT01599780
Title: On- and Off-line Measures of Language Development in Preterm Children
Brief Title: Language Development in Preterm Children
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Heidi M. Feldman, Professor, Stanford University
Other Study IDs: 18354
Record Dates: First submitted 2012-05-10; First posted 2012-05-16 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Language Development
Keywords: preterm; premature; prematurity; children; child; kid; toddler; infant; baby; language; development; skills; listening; talking; communication; speech; processing
MeSH Terms: conditions — Premature Birth; Deafness, Autosomal Recessive 1A; Language; Speech; Communication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Full-Term Children: ≥37 weeks gestation; 18 months old at the start of the study
- Preterm Children: <33 weeks gestation; 18 months old at the start of the study

SUMMARY:
This research investigates the ways in which preterm birth affects how very young children learn to speak and understand language, and how older children gain efficiency in language processing. The investigators observe how children at different ages learn new words and comprehend familiar words, how they communicate effectively with others, and how they use both linguistic and non-linguistic skills in problem-solving. All of the activities in the investigators' studies are designed to be age-appropriate and fun for children.

DETAILED DESCRIPTION:
In a typical session, the investigators video-record your child participating in one or more engaging activities with you and/or a member of the staff.

* In one type of task, your child looks at colorful pictures on a video screen while listening to recorded speech referring to the pictures. The investigators may vary factors in the speech stimuli such as word familiarity or sentence structure to learn more about the development of language understanding. Your child is seated on your lap throughout the session. From the video record, the investigators can later look at your child's gaze patterns in response to speech.
* In another type of task, the investigators observe children interacting with a staff member in the playroom. In these game-like activities, your child may be asked to play with toys, name or point to pictures, repeat sequences of words or sentences, tell stories, imitate hand movements, or solve puzzles. These observations help the investigators understand how language development relates to other types of cognitive activities in children at different ages.
* In a third type of task, the investigators observe how children interact spontaneously in a less structured situation. In some cases, the investigators observe you as you play with your child in a playroom. The investigators will provide you with a selection of toys appropriate to your child's age, and ask you to engage with your child as you would at home. From these observations, the investigators learn how children at different ages respond to language in the context of social interaction.

The investigators may also collect a language questionnaire and similar forms containing basic information about your child's development. Additionally, the investigators may review your child's medical records, including ultrasounds and MRI scans, to gain a better understanding of your child's medical history. All information is used for purposes of basic research on language learning only, and will not constitute a clinical assessment or evaluation.

TIME INVOLVEMENT

In this longitudinal study, each child is expected to come for a total of 12-16 sessions of behavioral testing, spread out over 3 years. Children are tested in 2 sessions (sessions occur approximately one week apart) at ages 18 (chronological), 18 (adjusted; applicable to pre-terms), 24, 30, 36, 42, 48, and 54 months. Each session typically lasts from 30 to 60 minutes, depending on the age of the child and number of breaks taken.

RISKS AND BENEFITS

There are no foreseeable risks or discomforts to you or your child in participating in this research. All the procedures are observational and non-intrusive. The investigators pace each session appropriately and give breaks as needed to enable your child to enjoy and complete the session. Your child will not be pressured to continue in the event that he or she becomes upset, tired, or resistant at any point during the session. If for any reason you or your child does not want to continue, the session will be ended immediately with no penalty.

The investigators cannot and do not guarantee or promise that you will receive any benefits from this study, apart from the payment and the satisfaction of participating in developmental research. If appropriate, the investigators provide information regarding resources that may be helpful in addressing any concerns regarding your child's development.

There are no direct costs to you for participating in this study. Neither you, nor your insurance provider, will be charged for the costs of any of the procedures performed for the purpose of this research study. The National Institute of Health is providing financial support for this study.

PARTICIPANT'S RIGHTS

If you have read this form and have decided to allow your child to participate in this project, please understand your child's participation is voluntary and your child has the right to withdraw his/her consent or discontinue participation at any time without penalty or loss of benefits to which he/she is otherwise entitled. Your child has the right to refuse to answer particular questions. The video record of the session will be identified by a code number, not by name. This record will be accessible only to the project directors and members of the project staff, unless you give your explicit permission for others to view it for scientific or educational purposes. All records will be stored securely so that your child's individual privacy will be maintained. In addition, your child's identity will remain private in all publications resulting from the study. Five years following the completion of your child's participation in this study, the investigators will destroy all raw videotapes.

ELIGIBILITY:
Inclusion Criteria:

* <33 weeks gestation
* <1800 grams at birth
* currently ≤ 18 months

Exclusion Criteria:

* an active seizure disorder (afebrile seizure within the last year) and/or anticonvulsant medication use
* central nervous system infections, revisions or other complications of a ventriculoperitoneal shunt for treatment for hydrocephalus, and/or congenital malformations
* history of a sensori-neural hearing loss, defined as 4-tone pure-tone average > 25 decibels
* visual impairments

Max Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born <33 weeks gestation (preterm)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
The Looking-While-Listening Task | 18 months, 18 months adjusted, 24 months, 30 months, & 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M Feldman, MD/PhD, Principal Investigator — Stanford University; Anne Fernald, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States